CLINICAL TRIAL: NCT06066034
Title: Changes in Serum, Follicular Fluid SREBP1c and LRG1 Levels in PCOS Patients and Correlation With Insulin Resistance
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gui Xiaoting (Other)
Responsible Party: Sponsor-Investigator, Gui Xiaoting, Resident physician, Zunyi Medical College
Organization: Zunyi Medical College (Other)
Other Study IDs: KLLY-2022-041
Record Dates: First submitted 2023-09-25; First posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: PCOS (Polycystic Ovary Syndrome) of Bilateral Ovaries
Keywords: PCOS; Insulin resistance
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Normal group: With the informed consent of the patient, venous blood was extracted on an empty stomach in the morning, and follicular fluid from multiple follicles was extracted during the 5-9 day menstrual cycle
- Insulin resistance group: With the informed consent of the patient, venous blood was extracted on an empty stomach in the morning, and follicular fluid from multiple follicles was extracted during the 5-9 day menstrual cycle
  Interventions: Diagnostic Test: HOMA-IR，ESHRE/ASRM
- PCOS group: With the informed consent of the patient, venous blood was extracted on an empty stomach in the morning, and follicular fluid from multiple follicles was extracted during the 5-9 day menstrual cycle
  Interventions: Diagnostic Test: HOMA-IR，ESHRE/ASRM
- PCOS with insulin resistance group: With the informed consent of the patient, venous blood was extracted on an empty stomach in the morning, and follicular fluid from multiple follicles was extracted during the 5-9 day menstrual cycle
  Interventions: Diagnostic Test: HOMA-IR，ESHRE/ASRM

INTERVENTIONS:
Diagnostic Test: HOMA-IR，ESHRE/ASRM — Grouping based on HOMA-IR and the diagnostic criteria of the European Society for Human Reproduction and Embryology and American Society for Reproductive Medicine (ESHRE/ASRM) in Rotterdam in 2003
  Groups: Insulin resistance group; PCOS group; PCOS with insulin resistance group

SUMMARY:
Polycystic ovary syndrome (PCOS) is a common reproductive endocrine and metabolic disease that affects 6-20% of women of childbearing age worldwide. Due to changes in modern lifestyles such as low fiber, high fat diets, sedentary lifestyles, smoking, and alcohol consumption, the risk of developing this disease has increased. Its clinical manifestations are heterogeneous, with typical clinical manifestations being oligomenorrhea or amenorrhea, infertility, hirsutism, and polycystic ovarian changes under ultrasound. Women affected by PCOS face significant reproductive challenges, seriously affecting their quality of life and increasing their psychological burden.LRG1 has various regulatory functions, including glucose and lipid metabolism, IR, angiogenesis, organ fibrosis, and inflammation. LRG1 can activate the transcription factor SREBP1 and participate in liver lipid synthesis in obese mice. SREBP1c is the active form of SREBP1. Research has shown that SREBP1c can directly or indirectly participate in the development of IR. Therefore, the investigators speculate that LRG1 may play a certain role in the progression of PCOS through SREBP1c.Understanding the local changes or metabolic characteristics of follicular fluid in patients with PCOS can help elucidate the pathogenesis of PCOS. Therefore, in this study,the investigators aim to detect changes in serum and follicular fluid LRG1, SREBP1c, and related hormone levels, and explore their role in the pathogenesis of PCOS from a systemic and ovarian perspective, providing new ideas for the prevention and treatment of PCOS and IR.

DETAILED DESCRIPTION:
1. The diagnostic criteria for all participants with polycystic ovary syndrome included in the study were based on the 2003 European Society for Human Reproductive and Embryonic Medicine and American Society for Reproductive Medicine (ESHRE/ASRM) diagnostic criteria in Rotterdam.
2. Collect basic data of all participants.
3. After informed consent, all participants were evaluated for insulin sensitivity(the degree of insulin resistance), using the insulin resistance index of the steady-state model. All participants were conducted after signing an informed consent form.
4. After informed consent, all participants were given fasting venous blood samples in the morning for measuring blood sugar, blood lipids, insulin, C-peptide, glycosylated hemoglobin (HbA1c), and a complete set of sex hormones.
5. After collecting follicular fluid from all participants, centrifuge at 1000xg for 20 minutes, filter and precipitate, and freeze in a refrigerator at -80 ° C for the determination of LRG1, SREBP1c, and related hormone levels in follicular fluid.
6. Use SPSS 22.0 statistical software for data analysis.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of Polycystic Ovary Syndrome

Exclusion Criteria:

Congenital adrenal cortical hyperplasia Adrenocortical carcinoma Cushing syndrome.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Sterile female
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Serum LRG1 levels | one years
  pg/ml
follicular fluid LRG1 levels | one years
  pg/ml
Serum SREBP1c levels | one years
  pmol/mL
follicular SREBP1c levels | one years
  pmol/mL

CONTACTS AND LOCATIONS:
Overall Officials: Fa Sun, Principal Investigator — Guizhou Provincial Health Commission
Locations (1):
- Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou, China